CLINICAL TRIAL: NCT03186924
Title: Reducing Sedentary Time in Rheumatoid Arthritis: The Take a STAND for Health Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Take a STAND for health RA
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Health

STUDY DESIGN:
Intervention Model Description: We will perform a 4-month parallel-group randomised controlled trial, in which rheumatoid arthritis patients will be assessed at baseline (PRE) and after 4 months (POST). Moreover, a sub-sample (n=18) of patients will perform a randomised crossover trial at baseline (PRE). Patients will complete three experimental sessions in a random manner, as follows: Prolonged sitting (SIT), in which participants engaged in prolonged sitting throughout an 8-h period and were instructed to minimize excessive movement; Exercise followed by prolonged sitting (EX), in which participants performed a 30-min moderate-to-vigorous exercise bout on a treadmill, subsequently, participants engaged in prolonged sitting as described for SIT; Light-intensity breaks (BR), in which participants completed a 3-min bout of light-intensity walking every 30 min of sitting throughout the experimental period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take a STAND for health (Experimental): A newly developed personalized intervention focused on replacing sedentary time with light-(or very light-) intensity physical activity
  Interventions: Behavioral: Take a STAND for health
- Control (No Intervention): The control group will receive all regular medical care and advice on healthy lifestyle, including the promotion of recommended physical activity levels and health nutrition.

INTERVENTIONS:
Behavioral: Take a STAND for health — The Take a STAND for health is a newly developed 4-month goal-setting intervention aimed at reducing sedentary behavior
  Arms: Take a STAND for health

SUMMARY:
This research program aims to comprehensively investigate the clinical, physiological, metabolic, and molecular effects of reducing sedentary behavior in rheumatoid arthritis. To this aim, we will conduct a 4-month parallel-group randomized controlled trial aiming to investigate the feasibility and efficacy of a newly developed personalized intervention focused on replacing sedentary time with light-(or very light-) intensity physical activity in rheumatoid arthritis. Additionally, a sub-sample of patients will complete a randomised cross-over study aiming to unravel potential mechanisms underlying the metabolic, physiological and molecular effects of breaking up sedentary time with light-intensity physical activity versus carrying out the minimum amount of daily exercise at once and then remaining sedentary versus simply remaining sedentary throughout all sessions, in a well-controlled laboratorial condition.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women diagnosed with rheumatoid arthritis

Exclusion Criteria:

* any physical disabilities that preclude physical exercise testing
* participation in structured exercise training programs within the last 12 months
* unstable dose of disease modifying drugs, including biological therapy, in the last 3 months prior to and during the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-12-17 (Estimated); Study Completion 2021-12-17 (Estimated)

PRIMARY OUTCOMES:
Sedentary behaviour as assessed by ActivPAL™ | 4 months

SECONDARY OUTCOMES:
Physical activity levels as assessed by ActiGraph GT3X® | 4 months
Disease activity as assessed by DAS28 | 4 months
Drug doses | 4 months
  Current and cumulative dose of prednisone, and current use of biological agents and non-biological disease-modifying anti-rheumatic drugs
Fatigue as assessed by the Fatigue Severity Scale | 4 months
Pain as assessed by the Visual Analogic Scale | 4 months (RCT) and 8 hours (crossover)
Body composition as assessed by densitometry (DEXA) | 4 months
  lean mass, fat mass and bone mass
Aerobic conditioning as assessed by a cardiopulmonary test | 4 months
Physical functioning as assessed by a Health Assessment Questionnaire | 4 months
Muscle function as assessed by a battery of tests | 4 months
  Timed Stands Test and Timed Up-and-Go Test
Blood pressure | 4 months (RCT) and 8 hours (crossover)
Insulin sensitivity as assessed by surrogates of insulin sensitivity | 4 months (RCT) and 8 hours (crossover)
  Glucose, insulin, c-peptide, and HbA1c
Inflammatory cytokines | 4 months (RCT) and 8 hours (crossover)
Lipid profile | 4 months (RCT) and 8 hours (crossover)
  Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides
Heart rate responses to exercise as assessed by a cardiopulmonary test | 4 months
  Chronotropic response and heart rate recovery
Muscle sympathetic nerve activity as assessed by microneurography | 4 months
Quality of life as assessed by the SF-36 questionnaire | 4 months
Western blotting | 4 months (RCT) and 8 hours (crossover)
RT-PCR | 4 months (RCT) and 8 hours (crossover)
RNA sequencing | 4 months (RCT) and 8 hours (crossover)
Lipidomics | 4 months (RCT) and 8 hours (crossover)
Vascular function and structure as assessed using a high-resolution ultrasound machine | 4 months
  Flow-mediated dilation and carotid intima-media thickness

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto AJ, Meireles K, Pecanha T, Mazzolani BC, Smaira FI, Rezende D, Benatti FB, DE Medeiros Ribeiro AC, DE Sa Pinto AL, Lima FR, Roschel H, Gualano B. Clinical and Cardiometabolic Effects of Reducing Sedentary Behavior in Postmenopausal Women with Rheumatoid Arthritis. Med Sci Sports Exerc. 2025 Jan 1;57(1):23-32. doi: 10.1249/MSS.0000000000003546. Epub 2024 Sep 16. PMID 39283176
- [Derived] Pinto AJ, Pecanha T, Meireles K, Benatti FB, Bonfiglioli K, de Sa Pinto AL, Lima FR, Pereira RMR, Irigoyen MCC, Turner JE, Kirwan JP, Owen N, Dunstan DW, Roschel H, Gualano B. A randomized controlled trial to reduce sedentary time in rheumatoid arthritis: protocol and rationale of the Take a STAND for Health study. Trials. 2020 Feb 12;21(1):171. doi: 10.1186/s13063-020-4104-y. PMID 32051025